CLINICAL TRIAL: NCT05340725
Title: The Population Pharmacokinetics and Pharmacodynamics of Rectal Dexmedetomidine Niosomes Administered for Postoperative Analgesia in Pediatric Cancer Patients.
Brief Title: Rectal Dexmedetomidine Niosomes for Postoperative Analgesia in Pediatric Cancer Patients.
Acronym: DEX-NANO
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hala Saad Abdel-Ghaffar, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SECI-IRB-IORG0006563
Record Dates: First submitted 2022-04-10; First posted 2022-04-22 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: This study will investigate the population pharmacokinetics and pharmacodynamics of rectal dexmedetomidine Niosomes for Postoperative Analgesia in Pediatric Cancer Patients undergoing bone marrow biopsy and aspiration in comparison with the intravenous and rectal plain formulation.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: An independent investigator not involved in the study will open the envelopes 1 h before induction of anesthesia and will prepare the study drug solutions in identical syringes and formulations with matching random codes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- DEX-IV (Active Comparator): Patients will receive iv DEX 1µ/kg diluted in 100 ml saline and given slowly iv infusion over 10 min. and rectal placebo 30 min. before induction of anesthesia.
  Interventions: Drug: DEX-IV
- DEX-Rectal (Active Comparator): Patients will receive rectal DEX suppository formulation at approximately 1µ/kg an iv. saline placebo. at 30 min. before induction of anesthesia.
  Interventions: Drug: DEX-Rectal
- DEX Nano-Rectal (Active Comparator): Patients will receive rectal DEX suppository in the Niosomes formulation at approximately 1µ/kg an iv. saline placebo at 30 min. before induction of anesthesia
  Interventions: Drug: DEX-Nano-Rectal

INTERVENTIONS:
Drug: DEX-IV — patients will receive iv DEX 1µ/kg diluted in 100 ml saline and given slowly iv infusion over 10 min. 30 min. before induction of anesthesia.
  Other Names: Precedex
  Arms: DEX-IV
Drug: DEX-Rectal — Patients will receive rectal DEX suppository formulation at approximately 1µ/kg at 30 min. before induction of anesthesia
  Other Names: Precedex
  Arms: DEX-Rectal
Drug: DEX-Nano-Rectal — Patients will receive rectal DEX suppository in the Niosomes formulation at approximately 1µ/kg at 30 min. before induction of anesthesia
  Other Names: Precedex
  Arms: DEX Nano-Rectal

SUMMARY:
Applying nanotechnology in drug delivery systems improved the bioavailability and kinetic profile of drugs in biological systems

DETAILED DESCRIPTION:
Nanotechnology which is focused on studying the properties and the applications of materials with structure size in the range of 1-100 nm has been widely used in various fields. In biomedical research fields, nanotechnology has been used to design and development of drug delivery systems (DDSs). Nanotechnology-based drug delivery systems (NDDSs) offer many potential advantages in cancer treatment, such as improving targeting of the therapeutic drugs, protecting drugs from degradation during in vivo transport, controlled drug release at specific sites or cells in response to specific signals, and thus improving the therapeutic efficacy while minimizing side effects.

Applying nanotechnology in drug delivery systems improved the bioavailability and kinetic profile of drugs in biological systems. Advances in nanotechnology aid in targeting drugs to specific molecular targets and safely delivering drugs to specific sites of action. The sustained release of nano-drug delivery systems enhances the controlled release profile of loaded drugs, thereby minimizing the dosage-regimen.

The aim of this study will be to investigate the population pharmacokinetics and pharmacodynamics of rectal dexmedetomidine Niosomes for Postoperative Analgesia in Pediatric Cancer Patients undergoing bone marrow biopsy and aspiration in comparison with the intravenous and rectal plain formulation.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I and II.
* Aged 3-7 yrs.
* Undergoing bone marrow aspiration and biopsy.

Exclusion Criteria:

* Allergy to the study drugs.
* Significant organ dysfunction.
* Cardiac dysrhythmia.
* Congenital heart disease.
* Use of psychotropic medication.
* Mental retardation.

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Serum concentrations of Dexmedetomidine | 6 hours.
  Pharmacokinetic parameters will be determined using noncompartmental method with WinNonlin professional Version 2.1 software (Pharsight Corporation, Mountain View, CA) based on measurement of plasma concentrations of DEX

SECONDARY OUTCOMES:
Postoperative FLACC pain score | 6 hours.
  Pain intensity will be assessed using the FLACC scale, with a maximum score of 10.

CONTACTS AND LOCATIONS:
Overall Officials: Hala Abdel-Ghaffar, MD, Principal Investigator — Professor of anesthesia and intensive care, faculty of medicine, Assiut university, Assiut, Egypt.
Locations (1):
- South Egypt cancer institute, Assiut university, Asyut, Assiut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No